CLINICAL TRIAL: NCT05384678
Title: Acute Dose-dependent Effects of DMT in Healthy Subjects: A Placebo-controlled Cross-over Study
Brief Title: Acute Dose-dependent Effects of DMT in Healthy Subjects
Acronym: DMT DR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2022-00378
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — N,N-Dimethyltryptamine

STUDY DESIGN:
Intervention Model Description: 5-period random order, placebo-controlled, double-blind cross-over study with four active substance conditions and placebo: 1. 0.6 mg/min, 2. 1.2 mg/min, 3. 1.8 mg/min, 4. 2.4 mg/min, 5. Placebo. Additionally, a patient-guided titration will be performed at the sixth and last session (not randomized).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- DMT 0.6 mg/min (Experimental)
  Interventions: Drug: N,N-Dimethyltryptamine (54 mg)
- DMT 1.2 mg/min (Experimental)
  Interventions: Drug: N,N-Dimethyltryptamine (108 mg)
- DMT 1.8 mg/min (Experimental)
  Interventions: Drug: N,N-Dimethyltryptamine (162 mg)
- DMT 2.4 mg/min (Experimental)
  Interventions: Drug: N,N-Dimethyltryptamine (216 mg)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- DMT 1.2 mg/min + dose titration (Experimental)
  Interventions: Drug: N,N-Dimethyltryptamine (108 mg) + dose titration

INTERVENTIONS:
Drug: N,N-Dimethyltryptamine (54 mg) — A dose rate of 0.6 mg/min will be administered
  Arms: DMT 0.6 mg/min
Drug: N,N-Dimethyltryptamine (108 mg) — A dose rate of 1.2 mg/min will be administered
  Arms: DMT 1.2 mg/min
Drug: N,N-Dimethyltryptamine (162 mg) — A dose rate of 1.8 mg/min will be administered
  Arms: DMT 1.8 mg/min
Drug: N,N-Dimethyltryptamine (216 mg) — A dose rate of 2.4 mg/min will be administered
  Arms: DMT 2.4 mg/min
Drug: Placebo — A Placebo (saline infusion) will be administered.
  Arms: Placebo
Drug: N,N-Dimethyltryptamine (108 mg) + dose titration — A dose rate of 1.2 mg/min will be administered with subsequent patient-guided dose titration
  Arms: DMT 1.2 mg/min + dose titration

SUMMARY:
N,N-dimethyltryptamine (DMT) is a psychoactive substance with similar effects such as LSD or psilocybin. However, DMT is less well characterized than the latter substances. The present study is a modern randomized cross-over trial, investigating different continuous intravenous DMT dose rates over a broad dose range. Thus, different doses will be tested and related to subjective and autonomic effects.

DETAILED DESCRIPTION:
N,N-dimethyltryptamine (DMT) is a naturally-occurring psychedelic substance widely used in recreational and spiritual settings (Ayahuasca). DMT is considered a tool to induce an altered state of consciousness of interest in psychological and psychiatric research. DMT is rapidly metabolized by monoamine oxidase (MAO) A. Therefore, it is inactive when administered orally and has a very short duration of action when administered parenterally (<20 min). In Ayahuasca, DMT is consumed together with harmala alkaloids that inhibit MAO to increase the oral bioavailablitity of DMT and to prolong its action after oral use. Alternatively, an intravenous administration regime including a bolus and maintenance perfusion has been proposed to induce a stable and prolonged DMT experience and is currently being investigated. However, to date no clinical study has investigated dose-response effects over a broad range of different doses of DMT within the same patient. The aim of the present study is to experimentally test different intravenous DMT doses over a broad dose range and investigate the related subjective and autonomic effects in order to establish a precise dose-response relationship of DMT in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years old
2. Sufficient understanding of the German language
3. Understanding of procedures and risks associated with the study
4. Willing to adhere to the protocol and signing of the consent form
5. Willing to refrain from the consumption of illicit psychoactive substances during the study
6. Abstaining from xanthine-based liquids from the evenings prior to the study sessions and during the sessions
7. Willing not to operate heavy machinery within 6 h of DMT administration
8. Willing to use double-barrier birth control throughout study participation
9. Body mass index between 18-29 kg/m2

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder (e.g. psychotic disorders, mania / hypomania, anxiety disorders).
3. Psychotic disorder or bipolar disorder in first-degree relatives
4. Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg)
5. Hallucinogenic substance use (not including cannabis) more than 20 times or any time within the previous two months
6. Pregnancy or current breastfeeding
7. Participation in another clinical trial (currently or within the last 30 days)
8. Use of medication that may interfere with the effects of the study medication
9. Tobacco smoking (>10 cigarettes/day)
10. Consumption of alcoholic beverages (>20 drinks/week)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Altered states of consciousness profile (5D-ASC) | 12 months
  5 Dimensions of Altered States of Consciousness (5D-ASC) consisting of 94 items to be rated on a visual analog scale (0-100 mm), with higher values indicating stronger effects with higher scores representing more intense effects.
  Assessed once on each study day
Subjective effect ratings over time | 12 months
  Participants will be asked by the investigator to repeatedly rate their subjective effects verbally on a Likert scale from 0 to 10 for: "any drug effect", "good drug effect", "bad drug effect", and "fear". Ratings will be performed before and repeatedly after substance administration and will take approximately 30 sec complete.

SECONDARY OUTCOMES:
States of consciousness questionnaire (SCQ) | 12 months
  Assesses the emergence and intensity of phenomenons occurring in altered states of consciousness on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely") once on each study day
Spiritual Realms Questionnaire | 12 months
  Assesses the spiritual phenomenons elicited by psychedelic substances through 11 main questions to be answered on a total of 65 sub-ordered 100mm visual analog scales once on each study day
Blood pressure | 12 months
  Assessed 20 times on each study day via systolic and diastolic blood pressure
heart rate | 12 months
  Assessed 20 times on each study day via heart rate
body temperature | 12 months
  Assessed 20 times on each study day via tympanic body temperature
Plasma level DMT | 12 months
  Assessed 22 times on each study day
Plasma level of oxytocin | 12 months
  Assessed 3 times on each study day
Plasma level of cortisol | 12 months
  Assessed 3 times on each study day
Plasma level of BDNF | 12 months
  Assessed 3 times on each study day
Plasma level of Prolactin | 12 months
  Assessed 3 times on each study day
Urine recovery of DMT | 12 months
  Assessed once on each study day
NEO-Five-Factor-Inventory (NEO-FFI) | Baseline
  The NEO-FFI is a self-description questionnaire with 60 items for the measurement of the "big five": neuroticism, extraversion, openness, agreeableness, and consciousness. It uses a 5-point Likert scale ranging from "completely disagree" to "fully agree".
Saarbrücker Personality Questionnaire (SPF) | Baseline
  The SPF defines empathy as the "reactions of one individual to the observed experiences of another." It assesses 28- items on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) each made up of 7 different items.
Elliot Humility Scale (EHS) | Baseline
  The Elliot Humility Scale (EHS) is a validated 13-item self-rating measure assessing four subscales, i.e. openness, self-forgetfulness, accurate self-assessment, and focus on others on a 5-point Likert scale ranging from "strongly disagree" to "strongly agree"

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, Principal Investigator — University Hospital Basel, Basel, Switzerland
Locations (1):
- Universtity Hospital Basel, Basel, Switzerland